CLINICAL TRIAL: NCT00585832
Title: Modifying Dietary Behavior in Adolescents With Elevated Blood Pressure
Acronym: DASH-4-Teens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Sarah C. Couch, Professor, University of Cincinnati
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: R01HL088567 (NIH); R01HL088567 (NIH)
Record Dates: First submitted 2007-12-27; First posted 2008-01-03 (Estimated); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Hypertension; Pre-Hypertension
Keywords: hypertension; pre-hypertension; adolescents; diet; vascular function
MeSH Terms: conditions — Hypertension; Prehypertension

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DASH-4-Teens Intervention (Experimental): DASH-4-Teens Intervention is described in detail in Couch, SC et al. Hypertension 2021: 77:241-251.
  Interventions: Behavioral: DASH-4-Teens
- Routine Care (Other): Routine Care is described in detail in Couch, SC et al. Hypertension 2021: 77:241-251.
  Interventions: Other: Routine Care

INTERVENTIONS:
Behavioral: DASH-4-Teens — 24-week behavioral nutrition intervention emphasizing a diet high in fruits, vegetables and low fat dairy foods and that is low in fat and sodium
  Arms: DASH-4-Teens Intervention
Other: Routine Care — individual in-person counseling sessions on guidelines consistent with the Fourth Pediatric Report of the National High Blood Pressure Education Program.
  Arms: Routine Care

SUMMARY:
The purpose of this study is to examine the long term effects of a 24-week clinically-based behavioral nutrition intervention emphasizing the DASH diet compared to routine nutrition care on changing diet quality, blood pressure, hypertension status, and vascular function in adolescents with elevated blood pressure.

DETAILED DESCRIPTION:
Hypertension in youth is no longer a rare disease and the number of affected children and adolescents is growing with the evolving pediatric epidemic in the US. Hypertension tracks from adolescence into adulthood and has been linked with preclinical indicators of adverse cardiovascular events in adults. Early prevention and intervention efforts are needed to address this increasing public and individual health problem. Preliminary studies from our research group demonstrate promising short-term effects of a behavioral nutrition intervention emphasizing a diet high in fruits, vegetables and low fat dairy that is also low in fat and sodium (the DASH diet) on lowering blood pressure (BP) in adolescents. The purpose of this application is to extend these findings by examining the long term effects of an improved 24-week clinically based behavioral nutrition intervention emphasizing the DASH diet (the DASH-4-Teens intervention) compared to routine nutrition care intervention on changing diet quality, BP, hypertension status, and vascular function in adolescents with elevated blood pressure. Adolescents with diagnosed pre-hypertension and stage 1 hypertension will be randomly assigned to receive either the DASH-4-teens intervention or routine nutrition care. The DASH-4- Teens intervention will include individual in-person nutrition counseling sessions, behavioral counseling telephone calls, and mailings. Routine nutrition care will include individual in-person counseling sessions on guidelines consistent with the Fourth Pediatric Report of the National High Blood Pressure Education Program. Primary outcomes will be measured in both conditions at 6 months (post-treatment) and at 1 year follow-up. Adherence to treatment will be measured as diet-related goals met, counseling session attendance, and telephone call and food monitoring completion. Findings are expected to improve the treatment of hypertensive adolescents in the clinical setting and contribute to the enhancement of the cardiovascular health of this population.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed pre-hypertension or stage 1 hypertension
* 11-18 years of age
* newly enrolled in the hypertension center at the Cincinnati Children's Hospital Medical Center

Exclusion Criteria:

* stage 2 hypertension
* secondary hypertension
* are being treated with anti-hypertensive medications
* have received prior formalized diet therapy to managed their blood pressure
* have target organ damage (as defined by a left ventricular mass index >51
* diagnosed type 1 or 2 diabetes
* use medications known to alter blood pressure
* are unwilling to stop use of vitamins, minerals or antacids
* do not speak English
* have a diagnosed eating disorder
* have a psychological or medical condition that may preclude them from full participation.
* do not have full medical clearance from a physician to participate

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 207 (Actual)
Dates: Start 2008-02; Primary Completion 2013-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Blood Pressure (BP) | change from baseline BP at immediately post-treatment (6 months)
  BP measurements were performed with a mercury sphygmomanometer according to standardized procedures. BP was calculated from the average of 2 BP measurements. Systolic and diastolic BP z-scores were made based on established norms.

SECONDARY OUTCOMES:
Vascular Function | change from baseline at immediately post-treatment (6 months)
  Flow mediated dilation (FMD) of the brachial artery was assessed using B-mode ultrasound vascular imaging according to Corretti MS et al., (J Am Coll Cardiology 2002; 39: 257-265).
DASH dietary adherence | change from baseline at immediately post-treatment (6 months)
  Dietary intake was assessed using 3 random 24 hour recalls (2 weekdays, 1 weekend day) collected in the 2 weeks before each assessment period using the validated multi-pass method. Recalls were collected from adolescents by telephone interview by trained dietitians using the Minnesota Nutrient Data Systems software (version 2.94, 2014). A DASH score was calculated according to Gunther et al (Hypertension 2009; 53: 6-12) modified to include a 10-point sodium component score. DASH score ranged from 0 to 90 with a higher score indicating greater DASH adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah C Couch, Ph.D., Principal Investigator — University of Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study are available from the corresponding author upon reasonable request.
Supporting Information: Study Protocol
Time Frame: through May 2023.
Access Criteria: The data that support the findings of this study are available from the corresponding author upon reasonable request.

REFERENCES:
- [Result] Couch SC, Saelens BE, Khoury PR, Dart KB, Hinn K, Mitsnefes MM, Daniels SR, Urbina EM. Dietary Approaches to Stop Hypertension Dietary Intervention Improves Blood Pressure and Vascular Health in Youth With Elevated Blood Pressure. Hypertension. 2021 Jan;77(1):241-251. doi: 10.1161/HYPERTENSIONAHA.120.16156. Epub 2020 Nov 16. PMID 33190559